CLINICAL TRIAL: NCT03573557
Title: Improved Intra-operative Safety From Optimal Selection of Anti-slip Surface
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE4817
Record Dates: First submitted 2018-06-15; First posted 2018-06-29 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Vaginal Surgery; Laparoscopic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pink Pad (Active Comparator): The Pink Pad will be used with subjects undergoing laparoscopic surgery or vaginal surgery while in to Trendelenburg to determine how much slipping is happening during the procedure.
  Interventions: Device: Pink Pad
- Bean Bag (Active Comparator): The Bean Bag will be used with subjects undergoing laparoscopic surgery or vaginal surgery while in to Trendelenburg to determine how much slipping is happening during the procedure.
  Interventions: Device: Bean Bag
- Gel Pad (Active Comparator): The Gel Pad will be used with subjects undergoing laparoscopic surgery or vaginal surgery while in to Trendelenburg determine how much slipping is happening during the procedure.
  Interventions: Device: Gel Pad

INTERVENTIONS:
Device: Pink Pad — Pink Pad made by Xodus Medical Inc. used for patients in steep Trendelenburg position during surgery.
  Arms: Pink Pad
Device: Bean Bag — Vac-Pac Bean Bag made by Olympic used for patients in steep Trendelenburg position during surgery.
  Arms: Bean Bag
Device: Gel Pad — Gel Pad used for patients in steep Trendelenburg position during surgery.
  Arms: Gel Pad

SUMMARY:
To identify the best surface to minimize the risk of intra-operative slipping when placed in Trendelenburg position. The outcomes of interest are to minimize the amount of movement from predefined anatomic landmarks and maximize the ease of performing the intended surgery. The study consists of performing a randomized trial comparing 3 common anti-slip surfaces to determine which surface provides the best result in terms of safety and cost.

DETAILED DESCRIPTION:
Laparoscopic surgery has become increasingly important in the drive to reduce patient morbidity. The introduction of robotic surgery has only served to accelerate this trend by allowing more complex surgeries to be performed using a minimally invasive technique. A key requirement of any minimally invasive gynecologic procedure is adequate visualization of the pelvis. This necessitates moving the bowel into the upper abdomen which is facilitated by placing patients in the Trendelenburg position. Steep Trendelenburg in the range of 30-40 degrees has historically been referenced as necessary for adequate visualization, but modern studies have found 16-28 degrees to be adequate. In practice, most physicians obtain the maximum Trendelenburg available as increasingly complex surgeries are attempted using minimally invasive techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo major laparoscopic or vaginal surgery by participating physicians at University Hospital Cleveland Medical Center
* Patients must not be pregnant

Exclusion Criteria:

* Pregnancy
* Patients unable to give consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 159 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Length of displacement when in Trendelenburg | 1 day
  Normal amount of displacement when place in Trendelenburg

SECONDARY OUTCOMES:
Cost of device | 1 day
  How cost effective is each surface
Rank of ease of use by physician | 1 day
  Surgeon will rate how the surface interferes with surgery
Number of adverse events | 1 day
  Count of adverse events per surface
Erythema score | 1 day
  Erythema score per surface graded by skin redness
Patient BMI | 1 day
  Influence of patient BMI on displacement per anti-slip surface
Patient age | 1 day
  Influence of patient age on displacement per anti-slip surface
Patient weight | 1 day
  Influence of patient weight on displacement per anti-slip surface
Patient height | 1 day
  Influence of patient height on displacement per anti-slip surface
Patient Hip circumference | 1 day
  Influence of patient hip circumference on displacement per anti-slip surface
Patient Waist circumference | 1 day
  Influence of patient waist circumference on displacement per anti-slip surface

CONTACTS AND LOCATIONS:
Overall Officials: Sherif El-Nashar, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States